CLINICAL TRIAL: NCT00601640
Title: Phase IIB Study to Evaluate the Safety and Efficacy of Topical Difluoromethylornithine and Topical Diclofenac in the Treatment of Sun-Damaged Skin on the Forearm
Brief Title: Eflornithine and/or Diclofenac in Treating Patients With Sun-Damaged Skin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-0032-04; P30CA023074 (NIH); P01CA027502 (NIH); UARIZ-BIO-06182 (Other: UA IRB no.); 07-0032-04 (Other: UA IRB)
Record Dates: First submitted 2008-01-22; First posted 2008-01-28 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: Other Benign Neoplasm of Skin, Unspecified
Keywords: skin cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — Diclofenac; Eflornithine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Eflornithine HCL (Experimental): Patients apply Eflornithine HCL ointment to their left forearm twice daily on days 1-90.
  Interventions: Drug: Eflornithine HCL ointment
- Diclofenac Na (Active Comparator): Patients apply topical Diclofenac Na gel to their left forearm once daily on days 1-90.
  Interventions: Drug: Diclofenac Na gel
- Eflornithine HCL and Diclofenac Na (Experimental): Eflornithine HCl ointment and Diclofenac Na gel applied twice and once daily, respectively on days 1-90.
  Interventions: Drug: Diclofenac Na gel; Drug: Eflornithine HCL ointment

INTERVENTIONS:
Drug: Diclofenac Na gel — Given topically twice daily on days 1-90
  Other Names: Solaraze
  Arms: Diclofenac Na; Eflornithine HCL and Diclofenac Na
Drug: Eflornithine HCL ointment — Given topically twice daily on days 1-90
  Other Names: Vaniqa
  Arms: Eflornithine HCL; Eflornithine HCL and Diclofenac Na

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. The use of eflornithine and diclofenac may stop cancer from growing in patients with sun-damaged skin.

PURPOSE: This randomized phase II trial is studying the side effects and how well eflornithine works compared with diclofenac, given alone or together, in treating patients with sun-damaged skin.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if combination therapy with topical eflornithine hydrochloride ointment and topical diclofenac sodium gel over 3-months increases the efficacy versus either agent used alone in the treatment of moderately sun-damaged skin.

Secondary

* To evaluate the safety of sequential administration of topical eflornithine hydrochloride ointment and topical diclofenac sodium gel.
* To determine the correlation of karyometric changes with histopathologic, immunohistochemical, clinical, and genetic polymorphism data.
* To obtain materials for microarray analysis.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

* Eflornithine hydrochloride : Patients apply topical eflornithine hydrochloride ointment to their left forearm twice daily on days 1-90.
* Diclofenac sodium : Patients apply topical diclofenac sodium gel to their left forearm once daily on days 1-90.
* Eflornithine hydrochloride/Diclofenac sodium : Patients apply topical eflornithine hydrochloride ointment as in arm I twice daily and topical diclofenac sodium gel as in arm II once daily on days 1-90.

Prior to treatment, three 4-mm punch biopsies are taken from the skin of the left lateral forearm for assessment of histopathology, the cyclooxygenase-2 enzyme and p53 expression, apoptosis, and nuclear chromatin karyometry. Tissue is also obtained for future use in microarray analysis. Blood is drawn for assessment of ornithine decarboxylase polymorphisms and for banking for subsequent studies. Biopsies are repeated 2-3 weeks after completion of treatment.

Digital photographs are taken at baseline and 1-2 weeks after completion of study therapy to document improvement of sun damage, appearance of new skin lesions, and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Visible sun-induced damage to the skin as assessed by the study dermatologists
* No inflammation of the skin on the lateral forearms
* No more than 10 actinic keratoses on the left forearm, and no actinic keratoses in the treatment area
* Resident of Pima or an adjoining Southern Arizona county
* History of treated basal cell carcinoma and/or squamous cell carcinoma of the skin at any site other than the left forearm allowed if excision or topical treatment was completed more than 30 days ago (60 days for radiotherapy)
* History of treated basal cell carcinoma and/or squamous cell carcinoma of the skin on the left forearm allowed 6 months after treatment is completed
* Must agree to avoid sun exposure to the left forearm as much as possible
* Not pregnant or nursing
* Not moderately to highly immunosuppressed by virtue of medication or disease, except for mildly suppressive disorders (e.g., diabetes mellitus or on mildly immunosuppressive therapy such as inhaled steroids for asthma)
* No serious concurrent illness that could interfere with study participation
* No active peptic ulcer disease, bleeding disorder, renal failure (creatinine > 2.0 mg/dL), or porphyria
* No known hypersensitivity to diclofenac sodium, eflornithine, acetylsalicylic acid, or NSAIDS
* No evidence of serious underlying medical conditions as demonstrated by abnormal values on baseline laboratory assessment
* More than 6 months since prior chemotherapy and in complete remission
* More than 60 days since prior and no concurrent oral diclofenac sodium (Cataflam®, Voltaren®, Voltaren-XR®) or combination of diclofenac and misoprostol (Arthrotec®)
* More than 60 days since prior and no concurrent IV eflornithine hydrochloride
* More than 30 days since prior and no concurrent topical retinoids, steroids, imiquimod (Aldara®), aminolevulinic acid HCl (Levulan®), eflornithine (Vaniqa®), diclofenac sodium gel (Solaraze®), or fluorouracil at any site
* More than 30 days since prior and no concurrent topical medication, other than emollients or sunscreens, on the left forearm
* Not undergoing concurrent bone marrow or solid organ transplant
* No concurrent immunosuppressive therapy (e.g., systemic chemotherapy or rheumatologic agents such as infliximab [Remicade®])
* No concurrent sunscreen use to the left forearm
* No concurrent active therapy for any invasive cancer
* No concurrent NSAIDs for more than 14 days per month for arthritic and other pain conditions
* Concurrent prednisone or other steroids with doses up to 20 mg/day (or the equivalent dose) allowed
* At least 30 days since prior and no concurrent enrollment on other investigational drug or device trial

Exclusion Criteria:

* Individuals receiving concurrent topical therapy with retinoids, steroids, 5-fluorouracil, Levulan, Vaniqa (eflornithine), Solaraze, or Imiquimod (Aldara®) within 30 days prior to study enrollment will be excluded. Subjects may be reconsidered for eligibility 30 days after the last topical treatment.
* Individuals who have had treatment for basal cell carcinoma or squamous cell carcinoma of the skin of the left forearm within six months prior to evaluation for the study will not be eligible. If interested, these subjects will be encouraged to return for re-evaluation once the six-month period is over.
* Individuals who are moderately to highly immunosuppressed by virtue of medication or disease will not be allowed to participate. This category includes individuals undergoing bone marrow or solid organ transplant, or receiving immunosuppressive therapy such as systemic chemotherapy or rheumatologic agents such as infliximab (Remicade®). However, individuals with mildly suppressive disorders such as diabetes mellitus or on mildly immunosuppressive therapy such as inhaled steroids for asthma will be eligible for participation. Doses up to 20 mg of prednisone per day or the equivalent dose of other steroids will be allowed.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2007-01; Primary Completion 2010-02 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M. Jeter, MD, Principal Investigator — University of Arizona
Locations (3):
- United States (3):
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare - Shea, Tucson, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona

REFERENCES:
- [Background] Bozzo P, Saboda K, Einspahr JG, Ranger-Moore J, Farmer ER, Cockerell CJ, Elder DE, Bangert JL, Hart N, Kramer CB, Alberts DS. Reliability and validity of a histologic score as a marker for skin cancer chemoprevention studies. Anal Quant Cytol Histol. 2003 Oct;25(5):285-92. PMID 14603727
- [Derived] Jeter JM, Curiel-Lewandrowski C, Stratton SP, Myrdal PB, Warneke JA, Einspahr JG, Bartels HG, Yozwiak M, Bermudez Y, Hu C, Bartels P, Alberts DS. Phase IIB Randomized Study of Topical Difluoromethylornithine and Topical Diclofenac on Sun-Damaged Skin of the Forearm. Cancer Prev Res (Phila). 2016 Feb;9(2):128-34. doi: 10.1158/1940-6207.CAPR-15-0232. Epub 2015 Dec 28. PMID 26712942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 184 participants were accrued. 18 were accrued when an interim analyses resulted in a change in formulation and dosing. The primary analyses is based on 166 accrued after this change.
Pre-assignment Details: 166 participants were accrued after the change in formulation. 10 participants were not randomized for various reasons. 156 participants were randomized to one of the 3 treatment groups.
Groups:
- Eflornithine Hydrochloride: Patients apply topical eflornithine hydrochloride ointment to their left forearm twice daily on days 1-90.
- Diclofenac Sodium: Patients apply topical diclofenac sodium gel to their left forearm once daily on days 1-90.
- Eflornithine Hydrochloride/Diclofenac Sodium: Patients apply topical Eflornithine hydrochloride ointment as in arm I twice daily and topical Diclofenac sodium gel as in arm II once daily on days 1-90.
Period: Overall Study
Arm/Group | Eflornithine Hydrochloride | Diclofenac Sodium | Eflornithine Hydrochloride/Diclofenac Sodium
Started | 52 | 52 | 52
Completed | 47 | 47 | 42
Not Completed | 5 | 5 | 10
Not completed — Withdrawal by Subject | 3 | 0 | 7
Not completed — Death | 1 | 0 | 0
Not completed — Adverse Event | 0 | 4 | 2
Not completed — intercurrent illness | 1 | 0 | 0
Not completed — change in eligibility status | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Patients apply topical eflornithine hydrochloride ointment to their left forearm twice daily on days 1-90.
- Arm II: Patients apply topical diclofenac sodium gel to their left forearm once daily on days 1-90.
- Arm III: Patients apply topical eflornithine hydrochloride ointment as in arm I twice daily and topical diclofenac sodium gel as in arm II once daily on days 1-90.
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Arm III | Total
Number analyzed (Participants) | 52 | 52 | 52 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 35 | 30 | 102
  >=65 years | 15 | 17 | 22 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (9.5) | 60.4 (11.0) | 61.4 (10.4) | 60.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 38 | 112
  Male | 15 | 15 | 14 | 44
Region of Enrollment [Number; unit: participants]
  United States | 52 | 52 | 52 | 156

OUTCOME MEASURES:

1. Primary Outcome: Changes in Putrescine Over 3 Months
Description: Putrescine is measured in nmole/g skin per biopsy. Baseline and End of Study biopsies were measured and the change was produced by subtracting baseline levels from End of Study levels. There was one baseline biopsy and one End of Study biopsy per participant.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: nmol/g skin
Arm/Group | Eflornithine Hydrochloride | Diclofenac Sodium | Eflornithine Hydrochloride/Diclofenac Sodium
Number analyzed (Participants) | 47 | 47 | 42
nmol/g skin | 0.03 (1.12) | 1.45 (1.23) | 0.2 (0.96)

2. Primary Outcome: Safety of Combination Therapy With Topical Eflornithine Hydrochloride Ointment and Topical Diclofenac Sodium Gel Over 3-months
Description: Adverse events were compared across three treatment groups by severity determined by the clinician. All adverse events were resolved by the end of follow up.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Eflornithine Hydrochloride | Diclofenac Sodium | Eflornithine Hydrochloride/Diclofenac Sodium
Number analyzed (Participants) | 52 | 52 | 52
participants
  Burning and Stinging None | 48 | 44 | 48
  Burning and stinging Mild | 4 | 8 | 3
  burning and stinging Moderate | 0 | 0 | 1
  Burning and Stinging Severe | 0 | 0 | 0
  Pruritis None | 42 | 33 | 40
  Pruritis Mild | 9 | 12 | 6
  Pruritis Moderate | 1 | 6 | 6
  Pruritis Severe | 0 | 1 | 0
  Rash, Redness. Erythema-None | 46 | 34 | 40
  Rash, Redness. Erythema-Mild | 5 | 10 | 7
  Rash, Redness. Erythema-Moderate | 1 | 8 | 5
  Rash, Redness. Erythema-Severe | 0 | 0 | 0
Statistical Analysis 1: Comparison: Eflornithine Hydrochloride vs Diclofenac Sodium vs Eflornithine Hydrochloride/Diclofenac Sodium; Test type: Superiority or Other; p = 0.022, Fisher Exact

3. Secondary Outcome: Change in Histologic Score Diagnosis and Treatment Group
Description: Change scores were computed by subtracting baseline histologic score from End of Study histologic score. Slides were formalin fixed. Histologic Score has been developed by this research group over the course of Grant (reference below). A standardized form captures data on the following criteria: basal or suprabasilar pleomorphism (atypia); inflammation; hyperkeratosis; parakeratosis. The atypia and inflammation were rated as: none (0), mild to moderate(1), and severe (2). The remaining criteria were rated as present (1) or absent (0). Histologic Scores were computed by adding together the codes for the histologic criteria. Higher scores reflected higher level of epidermal /dermal damage.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Eflornithine Hydrochloride | Diclofenac Sodium | Eflornithine Hydrochloride/Diclofenac Sodium
Number analyzed (Participants) | 48 | 46 | 42
units on a scale | 0.33 (0.15) | 0.26 (0.13) | 0.64 (0.18)

ADVERSE EVENTS:
Time Frame: Three months
Arm/Group | Arm I | Arm II | Arm III
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 20/52 | 45/52 | 28/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=52) | Arm II (N=52) | Arm III (N=52)
Burning/Stinging (Skin and subcutaneous tissue disorders) | 4 | 8 | 4
Rash, Redness, Erythema (Skin and subcutaneous tissue disorders) | 6 | 18 | 12
Pruritis (Skin and subcutaneous tissue disorders) | 10 | 20 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes